CLINICAL TRIAL: NCT05952037
Title: An Open-Label, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of the BCL2 Inhibitor Sonrotoclax (BGB-11417) as Monotherapy and in Combination With Zanubrutinib (BGB-3111) in Patients With Waldenström Macroglobulinemia
Brief Title: A Study to Investigate Efficacy and Safety of BCL2 Inhibitor Sonrotoclax as Monotherapy and in Combination With Zanubrutinib in Adults With Waldenström Macroglobulinemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-203; U1111-1291-4524 (Registry Identifier: World Health Organization); CTR20232718 (Registry Identifier: ChinaDrugTrials); 2023-503235-18-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Waldenstrom Macroglobulinemia; Waldenstrom's Macroglobulinemia Recurrent; Waldenstrom's Macroglobulinemia Refractory
Keywords: Waldenström's macroglobulinemia; Waldenstrom's Macroglobulinemia Recurrent; Waldenstrom's Macroglobulinemia Refractory; Lymphoma; BGB-11417; BCL-2i
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants with R/R disease to both Bruton tyrosine kinase (BTK) inhibitor and anti-CD20 antibody-based systemic therapy containing chemotherapy or proteasome inhibitor will receive sonrotoclax at a standard dose, given orally once daily.
  Interventions: Drug: Sonrotoclax
- Cohort 2 (Experimental): Participants with R/R disease to anti-CD20 antibody-based systemic therapy containing chemotherapy or proteasome inhibitor and were intolerant to BTK inhibitor will receive sonrotoclax at a standard dose, given orally once daily.
  Interventions: Drug: Sonrotoclax
- Cohort 3 (Experimental): Participants with R/R disease to a BTK inhibitor treatment and are unsuitable for chemoimmunotherapy will receive sonrotoclax at a standard dose, given orally once daily.
  Interventions: Drug: Sonrotoclax
- Cohort 4 (Experimental): Participants with previously untreated WM will receive sonrotoclax and zanubrutinib combination therapy for a fixed duration.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally as a tablet.
  Other Names: BGB-11417
Drug: Zanubrutinib — Administered orally as a capsule.
  Other Names: BRUKINSA; BGB-3111
  Arms: Cohort 4

SUMMARY:
This study will evaluate the safety and efficacy of the BCL2 inhibitor sonrotoclax (BGB-11417) in participants with relapsed/refractory Waldenström's Macroglobulinemia (R/R WM) and in combination with zanubrutinib in adult participants with previously untreated WM.

DETAILED DESCRIPTION:
This study will test whether sonrotoclax (BGB-11417) can be used to improve outcomes in participants with Waldenström's Macroglobulinemia (WM) both when used alone in those who have not responded well to conventional treatments and when used in combination with zanubrutinib in those who have not yet received treatment. The main goals of the study are to determine how many participants no longer have evidence of cancer or have some improvement in the signs and symptoms of cancer after treatment, and to determine what adverse events, or side effects, participants might experience.

BCL2 is a key protein involved in cell death, and abnormal levels of BCL2 are associated with many cancers. Blocking the action of BCL2 proteins is a promising approach with potential therapeutic benefits in participants with different types of cancers, including WM. This study will enroll approximately 105 participants. All participants will receive sonrotoclax orally as a tablet.

The study will take place at multiple centers worldwide. The overall time to participate in this study is approximately 5 years.

Note: Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and definitive histologic diagnosis of WM.
* Meeting ≥ 1 criterion for treatment according to consensus panel criteria from the 2nd International Workshop on Waldenström's Macroglobulinemia (IWWM).
* For Cohorts 1-3, refractory or relapsed disease at study entry unless participants had intolerance to the most recent therapy. Refractory disease is defined as not attaining at least a major response, or progressing while on or within 6 months of completing therapy. Relapsed disease is defined as attaining at least a major response to therapy and meeting the criteria for disease progression beyond 6 months after completing therapy.
* For Cohort 4, patients must not have received prior therapy for WM (except for plasmapheresis).
* Adequate organ function.

Exclusion Criteria:

* Central nervous system (CNS) involvement by WM.
* Transformation to aggressive lymphoma, such as diffuse large B-cell lymphoma.
* History of other malignancies ≤ 2 years before study entry.
* Uncontrolled active systemic infection or recent infection requiring parenteral antimicrobial therapy that was completed ≤ 14 days before the first dose of the study drug.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Major Response Rate (MRR) | Up to approximately 4 years
  MRR is defined as the percentage of participants achieving partial response (PR) or better, as assessed by the Independent Review Committee (IRC) per the 11th International Workshop on Waldenström Macroglobulinemia (IWWM-11) WM response criteria.

SECONDARY OUTCOMES:
Cohorts 2 and 3: MRR as assessed by the IRC | Up to approximately 5 years
  MRR is defined as the percentage of participants achieving PR or better.
All Cohorts: MRR as assessed by the Investigator | Up to approximately 5 years
  MRR is defined as the percentage of participants achieving PR or better.
Cohorts 1, 2, and 3: Duration of Major Response (DoMR) as assessed by the IRC | Up to approximately 5 years
  DoMR is defined as the time from first determination of major response until first documentation of progression or death, whichever occurs first.
All Cohorts: DoMR as assessed by the Investigator | Up to approximately 5 years
  DoMR is defined as the time from first determination of major response until first documentation of progression or death, whichever occurs first.
Cohorts 1, 2, and 3: Complete Response (CR) + Very Good Partial Response (VGPR) as assessed by the IRC | Up to approximately 5 years
  CR + VGPR is defined as the percentage of participants who achieve CR or VGPR.
All Cohorts: CR + VGPR as assessed by the Investigator | Up to approximately 5 years
  CR + VGPR is defined as the percentage of participants who achieve CR or VGPR.
Cohorts 1, 2, and 3: Overall Response Rate (ORR) as assessed by the IRC | Up to approximately 5 years
  ORR is defined as the percentage of participants with minor response (MR) or better.
All cohorts: ORR as assessed by the investigator | Up to approximately 5 years
  ORR is defined as the percentage of participants with MR or better.
Cohorts 1, 2, and 3: Duration of Response (DOR) as assessed by the IRC | Up to approximately 5 years
  DOR is defined as the time from first determination of response until first documentation of progression or death, whichever occurs first.
All Cohorts: DOR as assessed by the investigator | Up to approximately 5 years
  DOR is defined as the time from first determination of response until first documentation of progression or death, whichever occurs first.
Cohorts 1, 2, and 3: Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from first dose until first documentation of progression or death, whichever comes first, as assessed by the IRC and by the investigator.
Cohorts 1, 2, and 3: Time to major response as assessed by the IRC | Up to approximately 5 years
  Time to major response is defined as the time from start of study treatment to the first documentation of major response.
All Cohorts: Time to major response as assessed by the investigator | Up to approximately 5 years
  Time to major response is defined as the time from start of study treatment to the first documentation of major response.
Cohorts 1, 2, and 3: Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from first study drug administration to the date of death due to any cause.
Cohort 4: Time to next treatment | Up to approximately 5 years
  Defined as the time from the start of treatment to the start of first subsequent therapy for WM.
Number of participants reporting adverse events | Up to approximately 5 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory abnormalities, physical examination results, and vital signs.
All Cohorts: Change from Baseline in Health-Related Quality of Life (HRQoL): NFLymSI-18 Disease-related Symptoms-Physical and Treatment-Related Side Effects Subscales | Baseline and approximately months 7, 13, 19, and 25
  HRQoL based on participant-reported outcomes using National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Cancer Symptom Index - 18 Item (NFLymSI-18) Version 4. The questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and is divided into a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (72):
- United States (17):
  - City of Hope National Medical Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Northwestern Medicine Cancer Center, Warrenville, Illinois
  - Mission Cancer and Blood, Waukee, Iowa
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hattiesburg Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Atrium Health Levine Cancer Institute (Lci), Charlotte, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Ut Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Genesiscare North Shore, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Lions Gate Hospital Chemotherapy Clinic, North Vancouver, British Columbia
  - Qeii Health Science Center, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
- China (13):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Yancheng First Peoples Hospital, Yancheng, Jiangsu
  - Shengjing Hospital of China Medical Universityshenbei Branch, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University Branch South, Qingdao, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Third Peoples Hospital of Datong, Datong, Shanxi
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- France (6):
  - Centre Hospitalier Universitaire Damiens Hopital Sud, Amiens
  - Chu Clermont Ferrand Therapie Cellulaire and Hematolo, Clermontferrand
  - Institut Paoli Calmettes, Marseille
  - Hopital de La Pitie Salpetriere, Paris
  - Chu Hopital Lyon Sud, PierreBenite
  - Hopital Robert Debre, Reims
- General Hospital of Athens Alexandra, Athens, Greece
- Italy (7):
  - Irccs Azienda Ospedaliero Universitaria Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Istituto Europeo Di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Sanitaria Universitaria Friuli Centrale Presidio Ospedaliero Universitario Santa Maria Del, Udine
- Spain (7):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari Mutua Terrassa, Terrassa
- United Kingdom (9):
  - University Hospitals Dorset, Bournemouth
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - Nhs Highland, Inverness
  - St Jamess University Hospital, Leeds
  - University College Hospital, London
  - The Christie Nhs Foundation Trust Manchester, Manchester
  - Plymouth Hospitals Nhs Trust, Plymouth
  - Royal Marsden Nhs Foundation Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/